CLINICAL TRIAL: NCT01627951
Title: Comparison of NF54, NF135 and NF166 Strains of Plasmodium Falciparum in a Controlled Human Malaria Infection (TIP3)
Brief Title: Comparison of Three Plasmodium Falciparum Isolates in a Controlled Human Malaria Infection
Acronym: TIP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Havenziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TIP3
Record Dates: First submitted 2012-05-25; First posted 2012-06-26 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; malaria
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NF54 (Active Comparator): Volunteers will be infected with the NF54 strain of Plasmodium falciparum through the bites of 5 infected Anopheline mosquitoes.
  Interventions: Other: NF54
- NF135 (Experimental): Volunteers will be infected with the NF135 strain of Plasmodium falciparum through the bites of 5 infected Anopheline mosquitoes.
  Interventions: Other: NF135
- NF166 (Experimental): Volunteers will be infected with the NF166 strain of Plasmodium falciparum through the bites of 5 infected Anopheline mosquitoes.
  Interventions: Other: NF166

INTERVENTIONS:
Other: NF54 — Volunteers will be infected with the NF54 strain of Plasmodium falciparum through the bites of 5 infected Anopheline mosquitoes.
  Arms: NF54
Other: NF135 — Volunteers will be infected with the NF135 strain of Plasmodium falciparum through the bites of 5 infected Anopheline mosquitoes.
  Arms: NF135
Other: NF166 — Volunteers will be infected with the NF166 strain of Plasmodium falciparum through the bites of 5 infected Anopheline mosquitoes.
  Arms: NF166

SUMMARY:
An effective vaccine against malaria is urgently needed to combat the scourge of this disease. Before candidate vaccines can be tested in endemic countries, they are first tested in human volunteers in so-called Controlled Human Malaria Infections (CHMI's). Ideally, a candidate vaccine should be tested against multiple strains of malaria, representative of the disease's global distribution. To date, however, only one such strain (NF54) has been broadly used in CHMI's.

The purpose of this study is to compare the course of infections with 2 novel malaria strains to those with NF54 in human volunteers.

DETAILED DESCRIPTION:
Plasmodium falciparum (Pf) malaria remains responsible for an intolerable burden of morbidity worldwide and an effective vaccine is sorely needed to aid control efforts. Before candidate malaria vaccines can enter full-scale (phase IIb) field trials in endemic areas, they must first be tested under controlled circumstances in (phase IIa) clinical human malaria infection studies. Since Pf isolates display a wide genetic diversity across the globe, phase IIa challenge infections should be conducted with both homologous and heterologous strains.

Since 1998 a highly successful Controlled Human Malaria Infection model at the UMC St Radboud, Nijmegen, The Netherlands, has been employed both to test candidate vaccines and to answer fundamental questions about pathophysiological and immunological mechanisms during early Pf infection in human volunteers. To date largely the NF54 strain of P. falciparum has been used in this Nijmegen model, with which extensive experience has meanwhile been acquired. In order to increase the portfolio of Pf strains available for future phase IIa studies, it is first necessary to document in detail the parasitological, clinical and immunological characteristics of new candidate strains during a controlled human malaria infection. In this study, the strains NF135 and NF166 will be compared in this regard with the well-characterised NF54 strain.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 year-old healthy volunteers (males and females)
* General good health based on history,clinical examination and basic haematology and biochemistry results
* Negative pregnancy test in females
* Use of adequate contraception for females
* All volunteers must sign the informed consent form following proper understanding of the design and procedures of the study
* Volunteer agrees to inform his/her general practitioner and agrees to sign a request for medical information concerning possible contra-indications for participation in the study
* Willingness to undergo a Plasmodium falciparum sporozoite challenge
* Agreement to stay in a hotel room close to the trial center during a part of the study (day 5 post-infection until three days after initiation of treatment)
* Reachable by mobile phone during the whole study period
* Available to attend all study visits
* Agreement to refrain from blood donation to (Sanquin) blood bank or for other purposes, during the course of the study and for a minimum of three years thereafter
* Willingness to undergo an HIV, HBV and HCV test
* Negative urine toxicology screening test at screening visit and on the day before challenge
* Willingness to take a curative regimen of Malarone®

Exclusion Criteria:

* History of malaria
* Plans to travel to endemic malaria areas during the study period
* Previous participation in any malaria vaccine study and/or positive serology for P. falciparum
* Symptoms, physical signs and laboratory values suggestive of systemic disorders, including but not limited to renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the study results or compromise the health of the volunteer during infection
* History of diabetes mellitus or cancer (except basal cell carcinoma of the skin)
* Clinically significant ECG abnormalities at screening, or history of arrhythmia's or prolonged QT-interval
* Positive family history of cardiac disease in 1st or 2nd degree relatives <50 years old
* An estimated ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system
* Body Mass Index (BMI) below 18 or above 30kg/m2
* Any clinically significant deviation from the normal range in biochemistry or haematology blood tests or in urine analysis
* Positive HIV, HBV or HCV tests
* Participation in any other clinical study during or within 30 days prior to the onset of the trial
* Pregnant or lactating women
* Volunteers unable to give written informed consent
* Volunteers unable to be closely followed for social, geographic or psychological reasons
* Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the study
* A history of psychiatric disease or convulsions
* Known hypersensitivity to anti-malarial drugs
* History of severe reactions or allergy to mosquito bites
* The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months before study onset (inhaled and topical corticosteroids are allowed) or during the study period
* Contra-indications for Malarone® use including treatment taken by the volunteers that interfere with Malarone®
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including asplenia
* Co-workers of the department of Medical Microbiology of the UMC St Radboud or Havenziekenhuis, Rotterdam
* A history of sickle cell, thalassaemia trait and G6PD deficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Difference in kinetics of infection between groups infected with NF54, NF133 and NF166, as defined by a mathematical model that takes into account multiple measurements of parasitaemia | between day 5 and day 21
  Parasitaemia will be measured retrospectively by QRT-PCR in twice daily drawn venous whole blood, from day 5 post-infection until day of thick smear positivity, or else until day 21 post-infection if volunteers have not yet developed a positive thick smear before then. All these data points will be fed into a mathematical model that amalgamates them to calculate an outcome variable with one single value for burden of (liver-stage) infection and one for (blood-stage) multiplication factor.

SECONDARY OUTCOMES:
Difference in time till thick smear positivity between groups infected with NF54, NF135 and NF166 | between day 5 and day 21
  Thick smears will be read twice daily from day 5 post-infection until day of thick smear positivity, or else until day 21 post-infection
Difference in duration or peak height of parasitaemia between groups infected with NF54, NF135 and NF166 | between day 5 and day 21
  Parasitaemia will be measured retrospectively by QRT-PCR in twice daily drawn venous whole blood, from day 5 post-infection until day of thick smear positivity, or else until day 21 post-infection.
Difference in frequency of malaria-related symptoms and signs between groups infected with NF54, NF135 and NF166 | between day 5 and day 35
  Symptoms and signs will be assessed at twice daily check-up visits from day 5 post-infection until three days after thick smear positivity, or else until day 24 post-infection, and then again on day 35-post infection.
Difference in induced immunological responses between groups infection with NF54, NF135 and NF166 | between day -1 and day 35
  Peripheral venous whole blood will be drawn for assessment of serological and cellular immune responses on day 1-prior to infection, day 5 post-infection, day 9 post-infection and day 35 post-infection.

CONTACTS AND LOCATIONS:
Overall Officials: Perry van Genderen, MD PhD, Principal Investigator — Havenziekenhuis
Locations (2):
- Netherlands (2):
  - UMC St Radboud, Nijmegen
  - Havenziekenhuis, Rotterdam

REFERENCES:
- [Derived] McCall MBB, Wammes LJ, Langenberg MCC, van Gemert GJ, Walk J, Hermsen CC, Graumans W, Koelewijn R, Franetich JF, Chishimba S, Gerdsen M, Lorthiois A, van de Vegte M, Mazier D, Bijker EM, van Hellemond JJ, van Genderen PJJ, Sauerwein RW. Infectivity of Plasmodium falciparum sporozoites determines emerging parasitemia in infected volunteers. Sci Transl Med. 2017 Jun 21;9(395):eaag2490. doi: 10.1126/scitranslmed.aag2490. PMID 28637923